CLINICAL TRIAL: NCT07012304
Title: A Study on the Safety and Efficacy of Gecacitinib in Patients With Chronic Graft-versus-Host Disease (cGVHD) Who Have Received Prior Treatment With Two or More Systemic Therapies
Brief Title: Gecacitinib for cGVHD: Safety and Efficacy in Patients After ≥2 Lines of Prior Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yujun DONG (Other)
Responsible Party: Sponsor-Investigator, Yujun DONG, Director of the Hematology Department, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cGVHD-06
Record Dates: First submitted 2025-05-09; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: cGVHD; JAK inhibitor; Gecacitinib
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gecacitinib (Experimental)
  Interventions: Drug: Gecacitinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Gecacitinib Hydrochloride Tablets — Gecacitinib hydrochloride tablets are taken orally on an empty stomach. The starting dose is 50 mg once daily (QD). The maximum dose is 100 mg twice daily (BID), and the minimum dose is 50 mg every other day (QOD). Dose adjustments should be made in 50-mg increments or decrements.

SUMMARY:
Chronic Graft-versus-Host Disease (cGVHD) is a common late complication following allogeneic hematopoietic stem cell transplantation and a leading non-relapse cause of death. It is often treatment-refractory, significantly affecting patients' quality of life and prognosis. This study will evaluate the feasibility, safety, and tolerability of gecacitinib, a novel JAK and ACVR1 inhibitor, in 24 patients with moderate-to-severe cGVHD who have undergone two or more prior therapies. Participants will receive gecacitinib hydrochloride tablets for at least 24 weeks. Patients demonstrating disease stability, as assessed by the investigator, may continue treatment with the study drug until week 60, unless intolerability, disease progression, or initiation of new systemic therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily Signed informed consent and aged ≥18 years
* Undergone nonmyeloablative, myeloablative, or reduced-intensity allo-HSCT using bone marrow, peripheral blood stem cells, or umbilical cord blood from any donor source
* Confirmed myeloid and platelet engraftment: ANC >1.0×10⁹/L and platelet count >25×10⁹/L; no hematopoietic growth factors or blood product transfusions within 7 days before screening
* Clinically diagnosed moderate-to-severe cGVHD according to the 2014 NIH
* Received 2-5 prior systemic cGVHD therapies with persistent disease
* ECOG PS score of 0-2
* Able to swallow tablets
* Concomitant use of non-interacting immunosuppressants permitted

Exclusion Criteria:

* Recurrence of malignancy or loss of full donor chimerism
* Concurrent use of other JAK inhibitors, mesenchymal stem cells, or belumosudil (Eligible if discontinued for >8 weeks post-aGVHD treatment or stopped JAK inhibitors for cGVHD due to side effects.)
* Severe pulmonary cGVHD (FEV1 ≤39% or NIH lung symptom score of 3)
* Post-transplant lymphoproliferative disease
* Significant abnormalities affecting safety assessment, such as uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg) despite ≤2 antihypertensives; ALT/AST >3×ULN; DBIL/TBIL >1.5×ULN; serum creatinine >1.5×ULN
* History of major cardiovascular events within 6 months.
* Arrhythmia requiring treatment at screening
* Gastrointestinal conditions impairing drug absorption
* Surgery within 4 weeks of screening with incomplete recovery
* Active/uncontrolled infections (viral, bacterial, parasitic, fungal) requiring treatment
* Active tuberculosis within 6 months
* Epilepsy or use of psychotropic/sedative drugs
* Pregnant/breastfeeding or unwilling to use contraception during and 4 weeks post-study
* Malignancy within 5 years (except the indication for transplant)
* Use of anticoagulants/platelet inhibitors (except low-molecular-weight heparin)
* Herbal medicine use within 1 week prior to enrollment
* Hypersensitivity to gecacitinib or its components
* Participation in another clinical trial within 4 weeks (or 5 half-lives of the previous study drug, whichever is longer)
* Deemed unsuitable by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Week 24 | Week 24
  ORR was defined as the proportion of patients achieving complete response (CR) or partial response (PR) without requiring additional systemic therapy for cGVHD.

SECONDARY OUTCOMES:
ORR at Week 12, 48 and 60 | week 12, 48 and 60
Failure-free Survival (FFS) | Up to 24 months
Change From Baseline in Lee cGVHD Symptom Scale Scores | Through study completion, an average of 24 months
  Subscale scores and the summary score range from 0 to 100, with a higher score indicating worse symptoms.
Best Overall Response (BOR) | Up to week 24
Duration of Response (DOR) | Up to 24 months
Percentage of Participants With a ≥50% Reduction in Daily Corticosteroid Dose for ≥4 Weeks | Up to Day 180
Relapse Rate | Up to 24 months
Overall Survival (OS) | Up to 24 months
Change from Baseline in FACT-BMT | Through study completion, an average of 24 months
  The FACT-BMT (Functional Assessment of Cancer Therapy-Bone Marrow Transplant) total score ranges from 0 to 148. Higher scores reflect a better quality of life.
Change from Baseline in EQ-5D-5L | Through study completion, an average of 24 months
  The EQ-5D-5L (EuroQol 5-Dimension 5-Level Questionnaire) assesses health across five dimensions using five severity levels. It also includes a Visual Analogue Scale (VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health), where a higher score indicates a better health outcome.
Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | Up to 28 days after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China